CLINICAL TRIAL: NCT06915051
Title: Evaluation of the Relationship Between Umbilical Cord Coiling Index and Fetal Cardiac Functions.
Brief Title: The Relationship Between Umbilical Cord Coiling Index and Fetal Cardiac Functions.
Status: Completed | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEAH-COİLİNG
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Umbilical Cord Coiling Index and Fetal Cardiac Functions
Keywords: Umbilical cord coiling index; fetal cardiac functions; umbilical cord; fetal circulation
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This is a single-center study conducted on 200 randomly selected pregnant women with uncomplicated.
  Interventions: Diagnostic Test: Determining the relationship between the coiling number and fetal echocardiography findings.

INTERVENTIONS:
Diagnostic Test: Determining the relationship between the coiling number and fetal echocardiography findings. — Fetal echocardiography findings to be performed simultaneously with the determination of the coiling number.

SUMMARY:
The maximum efficiency of umbilical cord blood flow depends on a specific number of coils. With modern ultrasound techniques, investigators can now detect cord abnormalities even before birth. In recent years, there has been a renewed interest in the umbilical cord, and several articles have been published regarding the number of coils.In this study, the relationship between the umbilical cord coiling index and fetal cardiac functions was evaluated.

ELIGIBILITY:
Inclusion Criteria:

-Singleton uncomplicated pregnancies between 20-24 weeks seeking routine antenatal care.

Exclusion Criteria:

* Multiple pregnancy
* Preterm rupture of membranes
* Chorioamnionitis
* Placental abruption
* Severe fetal growth restriction
* Congenital anomalies of the fetus
* Preeclampsia
* Oligohydramnios
* Maternal diabetes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton uncomplicated pregnancies between 20-24 weeks seeking routine antenatal care will be included.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
The correlation between the fetal umbilical cord coiling number and the concurrently performed fetal echocardiography findings. | The correlation between the fetal umbilical cord coiling index and the echocardiographic findings of the fetus within the first hour will be investigated.
  This study will be a single-center study conducted on two hundred randomly selected pregnant women with uncomplicated singleton pregnancies in the late second trimester (20-24 weeks) who visit our hospital's perinatology outpatient clinic for routine prenatal check-ups. The umbilical cord coiling number and fetal cardiac function measurements will be performed within one hour by the same maternal-fetal medicine specialist.To optimize the quality of Doppler waveforms when assessing vascular structures, measurements will be obtained in the absence of uterine contractions and fetal activity, with an insonation angle as close to zero as possible and less than 30.Three parameters will be used to assess cardiac function:
  1. Diastolic function
  2. Systolic function
  3. Both systolic and diastolic function

CONTACTS AND LOCATIONS:
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No